CLINICAL TRIAL: NCT02460822
Title: Developing an mHealth Application to Improve Cancer Chemotherapy Symptom Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: McKesson Foundation (Other)
Responsible Party: Principal Investigator, Lawrence C. An, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-PAF07680
Record Dates: First submitted 2014-10-22; First posted 2015-06-02 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyChemoCare (Experimental): Participants will receive access to the the MyChemoCare iPad application, which allows them to track cancer and chemotherapy related symptoms daily, and suggests strategies that may help the participant deal with these symptoms. While using the application, high symptom severity scores will be reported to the participant's medical team, who may intervene to help relieve the symptom. Participants will also be contacted if they have not checked in for 48 hours to make sure they are coping well with their chemotherapy regimen.
  Interventions: Device: MyChemoCare iPad application

INTERVENTIONS:
Device: MyChemoCare iPad application

SUMMARY:
This research project addresses critical gaps in cancer symptom management through the creation of a mobile chemotherapy symptom management application. This application will assess for the presence and severity of common chemotherapy side-effects and provide personally tailored symptom-related video and narratives to enhance self-management of cancer and treatment-related symptoms. This study will examine patient acceptance and use of this mHealth application (called MyChemoCare) in a prospective trial of cancer patients (n=60) who are receiving chemotherapy for colorectal cancer at the University of Michigan Comprehensive Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colon or rectal cancer
* Expected to live at least 6 months
* Initiating chemotherapy for the first time in their treatment history
* Physically and mentally able to participate
* Able to read English
* Willing and able to sign informed consent

Exclusion Criteria:

* A treatment plan that does not include cytotoxic chemotherapy for colon or rectal cancer
* A medical history that includes cancer with the exception of in situ cancers of the cervix and basal cell cancers of the skin
* A current diagnosis that includes multiple cancers (this does not exclude metastatic disease)
* Received prior cytotoxic chemotherapy for any reason
* A diagnosed psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry C An, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MyChemoCare: Participants will receive access to the the MyChemoCare iPad application, which allows them to track cancer and chemotherapy related symptoms daily, and suggests strategies that may help the participant deal with these symptoms. While using the application, high symptom severity scores will be reported to the participant's medical team, who may intervene to help relieve the symptom. Participants will also be contacted if they have not checked in for 48 hours to make sure they are coping well with their chemotherapy regimen.
  MyChemoCare iPad application
Period: Overall Study
Arm/Group | MyChemoCare
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MyChemoCare
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Patient Retention and Engagement With the MyChemoCare Application
Description: Patient retention is defined as the number of patients who completed the 8-week study through the final evaluation. Engagement with the MyChemoCare application was measured as number of patients who checked in at least once per week of the study.
Time Frame: 8 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | MyChemoCare
Number analyzed (Participants) | 16
Participants
  Completed the 8-week trial | 15
  Checked in at least 1 time per week | 12

2. Primary Outcome: Patient Satisfaction and Usability of the MyChemoCare Application
Description: The investigators will use a 9-item survey developed by Dr. An to assess patients' experiences using the MyChemoCare app.
  This result is the mean of the the survey items (with opposite items reversed). The scale was scored from 0 = Strongly disagree to 6 = Strongly agree.
Time Frame: 8 weeks post enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MyChemoCare
Number analyzed (Participants) | 15
units on a scale | 3.95 (0.16)

3. Secondary Outcome: Physician Use of the Study Feedback Mechanism
Description: The investigators will assess for how many of the enrolled patients the physicians use the feedback from the app to assist in clinical care of the patients. This includes following up about distressing symptoms and using information provided by the patient during regular clinical visits.
Time Frame: 8 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | MyChemoCare
Number analyzed (Participants) | 16
Participants | 16

4. Secondary Outcome: Increased Mastery of Cancer and Chemotherapy Symptoms
Description: The investigators will use the Cancer Care Mastery Scale to assess patients' feelings of control over their cancer care. This scale is based on the Mastery Scale developed by Pearlin and Schooler, designed to capture the sense of control a patient feels over their cancer care. This is a 7-item scale where users are asked to respond to statements by choosing and answer from the following: Strongly disagree, Disagree, Neither agree or disagree, Agree, Strongly agree. Mastery scores were computed by taking the numeric mean of the items (1-5), with negatively worded items reversed.
  The number presented here is the number of patients whose mastery score improved between baseline and the end of the 8-week program. Because this is a small pilot study, we measure ANY improvement with no threshold specified.
Time Frame: 8 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | MyChemoCare
Number analyzed (Participants) | 15
Participants | 9

5. Secondary Outcome: Symptom Burden Reduction
Description: The investigators will use the MD Anderson Symptom Inventory (MDASI) to describe patient experiences in 8 core symptom areas (pain, fatigue, nausea, disturbed sleep, distress, lack of appetite, weakness, and diarrhea). For each area, patients are asked to rank their symptoms on a scale from 0 (Not present) to 10 (As bad as you can imagine). The overall score is the mean across all 8 items.
  The number reported here is the count of patients with a reduction in symptom burden between baseline and 8-week follow up. Because this is a small pilot study, we measure ANY reduction with no threshold specified.
Time Frame: 8 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | MyChemoCare
Number analyzed (Participants) | 15
Participants | 9

6. Secondary Outcome: Improved Quality of Life
Description: The investigators will use the FACT-G survey to assess four dimensions of patients health (physical, functional, social and emotional). For each of the dimensions, patients are given a series of statements about specific elements of well being and asked to rank them on the following scale: Not at all, a little bit, Somewhat, Quite a bit, or Very much. These items are given numeric values of 0-4, with negatively worded statements reverse coded. Within each of the four dimensions of health, average scores are calculated, and then an overall sum is derived. Total well-being ranges from 0 (Complete lack of well being) to 16 (Completely well).
  The number presented is the count of participants for whom the overall FACT-G score increased between baseline and 8-week followup. Because this is a small pilot study, we measure ANY increase with no threshold specified.
Time Frame: Baseline and 8 weeks post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | MyChemoCare
Number analyzed (Participants) | 15
Participants | 9

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | MyChemoCare
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
This was a feasibility pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No